CLINICAL TRIAL: NCT02405182
Title: Magnetic Resonance Imaging Biomarkers in Amyotrophic Lateral Sclerosis
Brief Title: MRI Biomarkers in ALS
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other); Western University, Canada (Other); McGill University (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Sanjay Kalra, Associate Professor, University of Alberta
Other Study IDs: RES0013831
Record Dates: First submitted 2015-02-27; First posted 2015-04-01 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS; Motor Neuron Diseases
Keywords: Magnetic Resonance Imaging; MRI; Biomarker
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: ALS patients (as well as patients with other motor neuron diseases such PLS and PMA) will be recruited from ALS clinics under the direction of ALS neurologists who are participating in this study. ALS patients should meet research criteria for possible, probable, probable laboratory-supported, or definite ALS. Patients with a history of CNS disease (e.g. stroke, head injury) or significant psychiatric disease will be ineligible. Patients must be able to undergo a brain MRI for approximately an hour.
  Interventions: Other: Magnetic Resonance Imaging
- Controls: Healthy controls who are age and gender matched to patients will be recruited. Controls with a history of CNS disease (e.g. stroke, head injury) or significant psychiatric disease will be ineligible. Controls must be able to undergo a brain MRI for approximately an hour.
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging
  Other Names: MRI

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a disabling and rapidly progressive neurodegenerative disorder. There is no treatment that significantly slows progression. Increasing age is an important risk factor for developing ALS; thus, the societal impact of this devastating disease will become more profound as the population ages. A significant hurdle to finding effective treatment has been an inability to accurately measure brain degeneration in humans. Advanced magnetic resonance imaging (MRI) techniques hold promise in this respect, and may assist in aiding diagnosis and the efficient testing of new drugs.

Different MRI features of brain degeneration will be measured in a large sample of patients with ALS. The study will operate within the Canadian ALS Neuroimaging Consortium (CALSNIC). CALSNIC is a clinical research platform comprised of ALS clinics with standardized clinical and neuroimaging protocols.

DETAILED DESCRIPTION:
This study will use advanced Magnetic Resonance Imaging (MRI) techniques to measure brain changes in ALS and related neurological conditions. Results from cognitive and neurological tests will be compared to the MRI. It is believed that these techniques will reveal changes in the brain that will help us understand normal brain function and the symptoms of neurological diseases as seen in ALS, as well to provide an objective measurement of degeneration (which is called a biomarker). This could improve not only the process by which new drugs for the treatment of neurological diseases are evaluated, but also how health care professionals address the needs of patients with these diseases.

Furthermore, a biomarker may give insight into the biological factors related to the diverse and variable clinical features amongst different patients.

Subjects will be recruited from ALS clinics that are a part of the Canadian ALS Neuroimaging Consortium (CALSNIC). Patients will have a diagnosis of ALS, PLS, PMA, or FTD. Healthy controls will be age and gender matched to patients. Subjects will visit their respective sites to undergo a clinical evaluation and an MRI. Follow up visits will occur at approximately 3-6 month intervals. Most subjects will have 2 follow up visits; more visits may occur for subjects who are physically able to continue in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be adults with a diagnosis of motor neuron disease (MND), including those with ALS, PLS, and PMA, and as well frontotemporal dementia (FTD) without motor neuron signs.
* Healthy controls over the age of 40 will also be recruited and will be age- and gender-matched to patients.

Exclusion Criteria:

* Subjects with other psychiatric/CNS illnesses such as Major Depressive Disorder, Schizophrenia, and Bipolar disorder, and those with significant head injury.
* Subjects ineligible for MRI investigation due to a pacemaker or other metallic foreign body, or significant claustrophobia that could affect the ability to have an MRI scan.

These exclusion criteria will also apply to controls.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited predominantly from ALS clinics at: the University of Alberta Hospital in Edmonton; the Foothills Medical Centre in Calgary; the Sunnybrook Health Sciences Centre in Toronto; the London Health Sciences Centre in London; and the Montreal Neurological Hospital in Montreal.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in neuronal and white matter integrity measures. | 24 months
  The primary analysis will evaluate changes in the brain using various advanced MRI techniques at baseline and specified follow up periods. Patients and controls scans will be compared.

SECONDARY OUTCOMES:
Correlation of neuronal and white matter integrity measures with clinical indices. | 30 months
  Secondary analyses will involve MRI comparison to clinical measures both at the time of the baseline scan and over time.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kalra, MD, FRCPC, Principal Investigator — University of Alberta
Locations (6):
- Canada (6):
  - University of Calgary / Heritage Medical Research Clinic, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia / GF Strong Rehab Centre, Vancouver, British Columbia
  - Western University / London Health Sciences Centre, London, Ontario
  - University of Toronto / Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University / Montreal Neurological Institute and Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Ta D, Ishaque A, Srivastava O, Hanstock C, Seres P, Eurich DT, Luk C, Briemberg H, Frayne R, Genge AL, Graham SJ, Korngut L, Zinman L, Kalra S. Progressive Neurochemical Abnormalities in Cognitive and Motor Subgroups of Amyotrophic Lateral Sclerosis: A Prospective Multicenter Study. Neurology. 2021 Aug 24;97(8):e803-e813. doi: 10.1212/WNL.0000000000012367. Epub 2021 Jun 14. PMID 34426551
- [Derived] Kalra S, Muller HP, Ishaque A, Zinman L, Korngut L, Genge A, Beaulieu C, Frayne R, Graham SJ, Kassubek J. A prospective harmonized multicenter DTI study of cerebral white matter degeneration in ALS. Neurology. 2020 Aug 25;95(8):e943-e952. doi: 10.1212/WNL.0000000000010235. Epub 2020 Jul 9. PMID 32646955